CLINICAL TRIAL: NCT03077711
Title: Methenamine Hippurate Versus Trimethoprim in the Prevention of Recurrent UTIs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Carolyn Botros, Female Pelvic Medicine and Reconstructive Surgery, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EH16-216
Record Dates: First submitted 2017-02-27; First posted 2017-03-13 (Actual); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Urinary Tract Infections, Recurrent
MeSH Terms: conditions — Urinary Tract Infections | interventions — Trimethoprim; methenamine hippurate

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with recurrent urinary tract infections are recruited into this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with recurrent UTIs arm 1 (Active Comparator): Patients are randomized to receive methenamine hippurate in one arm if they are diagnosed with recurrent urinary tract infections.
  Interventions: Drug: Methenamine hippurate
- Patients with recurrent UTIs arm 2 (Active Comparator): Patients are randomized to receive trimethoprim in the other arm if they are diagnosed with recurrent urinary tract infections.
  Interventions: Drug: Trimethoprim

INTERVENTIONS:
Drug: Trimethoprim — suppressive antibiotic. Estrogen cream may be prescribed if the patient is post-menopausal (but not as a part of this study).
  Other Names: Trimpex
  Arms: Patients with recurrent UTIs arm 2
Drug: Methenamine hippurate — antiseptic used in the prevention of recurrent UTIs. Estrogen cream may be prescribed if the patient is post-menopausal (but not as a part of this study).
  Other Names: Hiprex
  Arms: Patients with recurrent UTIs arm 1

SUMMARY:
Several methods are available for use in the prevention of recurrent urinary tract infections (UTIs) over the past few decades. These methods include suppressive antibiotics, estrogen cream, methenamine hippurate, d-mannose, cranberry, probiotics, and vitamin C. Of these, the majority of the literature is in favor of use of suppressive antibiotics for preventing UTIs. However, this data is now about 10 years old. Increasing use of antibiotics over the years has lead to increased resistance of bacteria. In addition, long-term antibiotic use has several adverse effects, some life-threatening. There is recent literature evaluating the use of several of the alternatives to suppressive antibiotics with mixed results. A comparative study of the efficacy of methenamine hippurate to suppressive antibiotics is lacking in the current literature. Several early partly-randomized trials done with methenamine hippurate have shown promising results, but are only as recent as 1987. The primary objective of this prospective, randomized study is to determine whether there is a significant difference in the prevention of recurrent UTIs when given either methenamine hippurate or daily suppressive antibiotics. The secondary objective of this study is to determine how well patients are able to tolerate each of these medications and what adverse effects are observed in a given 1 year time period. The long-term goals of this study are to find an alternative to using suppressive antibiotics, potentially with a lower adverse effect profile and less of the dangers of long term antibiotic use. Finding an alternative to suppressive antibiotics would also tackle the issue of antibiotic resistance.

DETAILED DESCRIPTION:
Hypothesis:

The hypothesis of this study is that the group taking trimethoprim will have a lower recurrence rate than those taking methenamine hippurate based on the literature. The investigators aim to identify to what degree that difference is and whether or not it is an acceptable difference given the greater degree of an antibiotic resistance.

Objectives:

The primary objective of this prospective, randomized study is to determine whether there is a significant difference in the prevention of recurrent UTIs when given either methenamine hippurate or daily suppressive antibiotics independent of vaginal estrogen use.

The secondary objective of this study is to determine how well patients are able to tolerate each of these medications and what adverse effects are observed in a 1 year time period.

Specific Aims:

1. Identify if there is a differential impact on prevention of recurrent UTIs when treated with either trimethoprim or methenamine hippurate in a 6 and 12 month period.
2. Identify adverse reactions in each group.
3. Determine whether or not estrogen has a more additive effect to trimethoprim or methenamine hippurate in post-menopausal women.
4. Identify how well tolerated the study medications are and whether or not the size of the pills or the frequency of taking them prevents patients from continuing therapy.

ELIGIBILITY:
Inclusion Criteria:

* recurrent UTI: at least 2 in the past 6 months or 3 in past year (culture positive)
* must have been symptomatic with dysuria, urgency, frequency, suprapubic pain, hematuria, malodorous urine
* treated for last UTI and negative urine culture on entry into study
* English speaking

Exclusion Criteria:

* pregnancy
* urinary tract abnormalities (eg kidney stones)
* acute pyelonephritis
* renal insufficiency or failure
* known allergy to medications
* prophylaxis for post-coital recurrent UTIs

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore Univeristy HealthSystem, Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The investigators are currently only recruiting at one institution and only researchers on the original institutional review board will have access to data. Only the principal investigator and research coordinator will have the data to be analyzed.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 104 patients actually signed consent to participate but 12 were excluded due to screening failure, decision to decline participation after signing consent, renal failure discovered after enrolling patient, and one unrelated death
Groups:
- Patients With Recurrent UTIs Arm 1: Patients are randomized to receive methenamine hippurate in one arm if they are diagnosed with recurrent urinary tract infections.
  Methenamine hippurate: antiseptic used in the prevention of recurrent urinary tract infections (UTIs).
- Patients With Recurrent UTIs Arm 2: Patients are randomized to receive trimethoprim in the other arm if they are diagnosed with recurrent urinary tract infections (UTIs).
  Trimethoprim: suppressive antibiotic.
Period: Overall Study
Arm/Group | Patients With Recurrent UTIs Arm 1 | Patients With Recurrent UTIs Arm 2
Started | 47 | 45
Completed | 43 | 43
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — noncompliant taking medication | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Recurrent UTIs Arm 1 | Patients With Recurrent UTIs Arm 2 | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (15.4) | 73 (10.5) | 72 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 45 | 92
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 45 | 92
BMI [Mean (Standard Deviation); unit: kg/m2] | 30 (6.4) | 30 (7.7) | 30 (6.9)
Parity [Mean (Standard Deviation); unit: number of births] | 2.7 (2.2) | 2.3 (1.4) | 2.5 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Time to Subsequent Infection as Defined From Time of Treatment Initiation to Recurrence of UTI
Description: Patients will be advised to follow up with any symptoms of a recurrence or at 6 and 12 month intervals if symptom-free.
Time Frame: up to 12 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- Patients With Recurrent UTIs Arm 1: Patients are randomized to receive methenamine hippurate in one arm if they are diagnosed with recurrent urinary tract infections.
  Methenamine hippurate: antiseptic used in the prevention of recurrent UTIs.
- Patients With Recurrent UTIs Arm 2: Patients are randomized to receive trimethoprim in the other arm if they are diagnosed with recurrent urinary tract infections.
  Trimethoprim: suppressive antibiotic.
Arm/Group | Patients With Recurrent UTIs Arm 1 | Patients With Recurrent UTIs Arm 2
Number analyzed (Participants) | 43 | 43
days | 101 (84.4) | 119 (94)

2. Primary Outcome: Recurrent UTI
Description: The number of patient who had a recurrence of UTI within 12 months
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Recurrent UTIs Arm 1 | Patients With Recurrent UTIs Arm 2
Number analyzed (Participants) | 43 | 43
Participants | 28 | 28

3. Primary Outcome: Number of Infections
Description: The number of infections at a 12 month follow up time period as defined by symptoms and positive urine culture.
Time Frame: up to 12 months
Measure: Mean (Standard Deviation); unit: urinary tract infections
Arm/Group | Patients With Recurrent UTIs Arm 1 | Patients With Recurrent UTIs Arm 2
Number analyzed (Participants) | 43 | 43
urinary tract infections | 1.5 (1.7) | 1.6 (1.9)

4. Secondary Outcome: Adverse Effects
Description: The percentage of patients complaining of adverse effects of each medication, including dyspepsia, dysuria, rash, pruritus, nausea, epigastric pain, vomiting, glossitis, taste changes, fever, and photosensitivity.
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Recurrent UTIs Arm 1 | Patients With Recurrent UTIs Arm 2
Number analyzed (Participants) | 47 | 45
Participants
  diarrhea | 1 | 2
  rash | 2 | 0
  clostridium difficele infection | 1 | 0
  weakness | 2 | 0
  abdominal pain | 0 | 1
  kidney stone | 0 | 1
  no adverse event | 41 | 41

5. Secondary Outcome: Morisky Medication Adherence Survey
Description: Morisky Medication Adherence Scale-8 (MMAS-8). Patient tolerability of medications using a tolerability survey. Minimum and maximum scores are 0 and 8 respectively. 0 means no adherence and 8 is maximal adherence. Low adherence corresponds to a score less than 6, medium adherence is between 6 and <8, and 8 is high adherence.
Time Frame: up to 12 months
Population: We were not able to obtain the Morisky medication survey on all participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients With Recurrent UTIs Arm 1 | Patients With Recurrent UTIs Arm 2
Number analyzed (Participants) | 30 | 21
units on a scale | 7.28 (1.1) | 6.94 (1.6)

6. Secondary Outcome: Bacterial Infection Prevalence and Types
Description: Urine cultures and sensitivities for positive urine cultures
Time Frame: up to 12 months
Measure: Number; unit: infections
Arm/Group | Patients With Recurrent UTIs Arm 1 | Patients With Recurrent UTIs Arm 2
Number analyzed (Participants) | 47 | 45
infections
  Escherichia coli | 43 | 50
  Klebsiella pneumonia | 11 | 6
  Enterococcus faecalis | 3 | 9
  Extended spectrum beta lactamase Escherichia coli | 6 | 9
  Other bacteria | 15 | 12
  Strains pan sensitive to all antibiotics | 5 | 20
  Strains resistant to trimethoprim | 58 | 30
  Strains resistant to abx other than trimethoprim | 10 | 29

ADVERSE EVENTS:
Time Frame: Over 1 year from entry into the study
Arm/Group | Patients With Recurrent UTIs Arm 1 | Patients With Recurrent UTIs Arm 2
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/45
Other Adverse Events (participants affected / at risk) | 6/47 | 4/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Recurrent UTIs Arm 1 (N=47) | Patients With Recurrent UTIs Arm 2 (N=45)
diarrhea (Gastrointestinal disorders) | 1 | 2
rash (Skin and subcutaneous tissue disorders) | 2 | 0
clostridium difficele colitis (Gastrointestinal disorders) | 1 | 0
weakness (General disorders) | 2 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 1
kidney stone (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT03077711/Prot_SAP_000.pdf